CLINICAL TRIAL: NCT00507897
Title: Hemodynamic Parameters in Euthyroid Patients With Thyroid Nodules
Status: Terminated | Type: Observational
Why Stopped: The received reliability with increase in quantity of participants of research did not vary
Sponsor: Yaroslavl State Medical Academy (Other)
Other Study IDs: ESheverdova-1
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-02

CONDITIONS: Thyroid Nodules
Keywords: thyroid nodules, blood pressure, thyroid hormones
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: Cohort: Patients with normal blood pressure scheduled to have thyroid nodules surgically removed
- A1: Patients from group A not receiving any drugs and who lack other pathology, gender and age matched group B1
- B: Cohort: Patients with increased blood pressure scheduled to have thyroid nodules surgically removed
- B1: Patients from group B not receiving any drugs and who lack other pathology, gender and age matched group A1

SUMMARY:
The purpose of this study is to determine the relationship of hemodynamic parameters with the level of thyroid hormones and the histological structure of thyroid nodules in euthyroid patients.

DETAILED DESCRIPTION:
As opposed to widely investigated condition of cardiovascular system in patients with functional disorders of thyroid gland, the relationship between thyroid hormones and hemodynamic parameters in euthyroid patients remains not enough clear.

We detect the parameters of blood pressure and thyroid hormones in euthyroid patients with thyroid nodules directly before planned operation on the thyroid gland.

As the study is carries out directly before operation, that assumes presence of preoperative stress in patients, activity of the sympatho - adrenal system is estimated in addition.

On the one hand, the design of our research will allow to estimate relationship of thyroid hormones with the parameters of blood pressure in conditions of euthyroidism, on the other hand - to investigate features of blood pressure in patients with thyroid nodules.

The research of the patients in the preoperative period will enable to select the group of patients without pathology of cardiovascular system whose increased blood pressure is connected with preoperative stress, that in turn will allow to exclude influence of the pathology of the cardiovascular system on studied correlation.

ELIGIBILITY:
Inclusion Criteria:

* Euthyroid patients with thyroid nodules before operation on the thyroid gland

Exclusion Criteria:

* Hyperthyroidism
* Hypothyroidism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Alexandrov, Professor, Study Chair — Yaroslavl State Medical Academy
Locations (1):
- Yaroslavl State Medical Academy, Yaroslavl, Russia